CLINICAL TRIAL: NCT03608111
Title: Effects of Single-task Versus Dual-task Training on Balance Performance in Elderly Osteoarthritic Patients With Balance Impairment
Brief Title: Effects of Single-task Versus Dual-task Training on balancePERFORMANCE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ufuk University (Other)
Responsible Party: Principal Investigator, ASLIHAN UZUNKULAOGLU, Ufuk University, Ufuk University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 30112015-5.
Record Dates: First submitted 2018-07-23; First posted 2018-07-31 (Actual); Last update posted 2018-07-31 (Actual); Status verified 2018-07

CONDITIONS: Balance Impairment

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- single task balance training (Active Comparator)
  Interventions: Other: single task balance training; Other: dual task balance training
- dual task balance training (Active Comparator)
  Interventions: Other: single task balance training; Other: dual task balance training

INTERVENTIONS:
Other: single task balance training — single task balance training
Other: dual task balance training — dual task balance training

SUMMARY:
Background: Impairment in the control of balance is a common problem among elderly patients especially whom with osteoarthritis (OA).

Aim: The aim of this study was to compare the effects of single-task and dual-task training on balance performance in the elderly osteoarthritic patients with balance impairment.

DETAILED DESCRIPTION:
Fifty elderly osteoarthritic patients with balance impairment were included into this study. Patients were randomly assigned to single task balance training (Group 1) or dual-task balance training (Group 2) groups. Balance activities were given to both groups for 3 times a week for 4 weeks. Patients in group 2 also performed cognitive tasks simultaneously with these exercises. Patients were evaluated with Berg balance scale (BBS), kinesthetic ability trainer (KAT 2000) static and dynamic scores, timed up and go test (TUTG) and walking speed for single and dual tasks, number of stopping and Activities Specific Balance Confidence (ABC) Scale at the baseline and at the end of 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* included age ≥65, able to walk 10 m, no neurological or musculoskeletal diagnosis, met the criteria of balance impairment, and scored >19 on the mini mental state examination.

Exclusion Criteria:

* neurologic or musculoskeletal diagnosis such as stroke, orthopedic involvement, significant visual and auditory impairments, severe vitamin B12 deficiency and sedative drug use.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2017-01-01 (Actual); Study Completion 2017-01-01 (Actual)

PRIMARY OUTCOMES:
Berg balance scale | 1 month

IPD SHARING:
Plan to Share IPD: No